CLINICAL TRIAL: NCT02924181
Title: Comparison of Acute Pulmonary Vein (PV) Reconnection Between Contact Force Guided and Blinded PV Isolation in Patients With Symptomatic Atrial Fibrillation
Brief Title: Comparison Between Contact Force Guided and Blinded Strategy on PV Isolation in AF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH
Record Dates: First submitted 2016-05-19; First posted 2016-10-05 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein isolation; contact force sensing catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lt PV CF guided/rt PV CF blinded (Active Comparator): Fifteen patients will be allocated to this group. Left side pulmonary veins isolation will be performed with contact force information guidance. Then, right side pulmonary veins isolation will be performed without contact force information (using same catheter named SmartTouch Catheter).
  Interventions: Device: SmartTouch Catheter
- Lt PV CF blinded/rt PV CF guided (Active Comparator): Fifteen patients will be allocated to this group. Left side pulmonary veins isolation will be performed without contact force information (using same catheter named SmartTouch Catheter).Then, right side pulmonary veins isolation will be performed with contact force information guidance.
  Interventions: Device: SmartTouch Catheter
- Rt PV CF guided/lt PV CF blinded (Active Comparator): Fifteen patients will be allocated to this group. Right side pulmonary veins isolation will be performed with contact force information guidance. Then, left side pulmonary veins isolation will be performed without contact force information (using same catheter named SmartTouch Catheter).
  Interventions: Device: SmartTouch Catheter
- Rt PV CF blinded/lt PV CF guided (Active Comparator): Fifteen patients will be allocated to this group. Right side pulmonary veins isolation will be performed without contact force information (using same catheter named SmartTouch Catheter). Then, left side pulmonary veins isolation will be performed with contact force information guidance.
  Interventions: Device: SmartTouch Catheter

INTERVENTIONS:
Device: SmartTouch Catheter — Pulmonary vein (PV) isolation guided by CF information
  Other Names: Contact force guided pulmonary vein isolation

SUMMARY:
Pulmonary vein (PV) isolation is very important in atrial fibrillation (AF) catheter ablation. PV reconnection is one of the main reasons in AF recurrence. Contact force-sensing catheter is a new catheter which has valuable tools to monitor and increase the efficacy of PV isolation. Previous paper reported the efficacy of contact force-sensing catheter on immediate PV isolation and outcome. However, there might be confounding factor as inter-individual variation. Therefore, we would like to compare the efficacy of contact force-sensing catheter within same patient but different veins.

In this study, we would like to confirm the efficacy of contact force-sensing catheter on immediate PV isolation outcome within same patient. This study randomized the right or left PVs whether to use the contact force-sensing function or not. The study design will minimize the inter-individual variation on evaluating the efficacy of contact force-sensing catheter on immediate PV isolation.

Also, in patients who had recurred AF or AT, we would like to evaluate the long-term efficacy of contact force-sensing catheter on PV isolation.

DETAILED DESCRIPTION:
Sixty patients will be randomized to select right or left pulmonary veins whether to apply contact force-guided ablation or contact force-blinded ablation strategy. Each PV will be ablated with same contact force-sensing catheter (Thermocool Smart Touch Catheter, Biosense Webster Inc. CA). The PV (right or left) which will be randomized to contact force-sensing PV or blind PV. Contact force-sensing PV will be ablated guided by contact force, whereas the blind PVs will be ablated without contact force-sensing information. The change of impedance, total ablation and time to ablate PV will be collected and analysed according to contact force-sensing strategy. After exit and entrance block by conventional method, dormant conduction will be evaluated by using adenosine. The proportion of dormant conduction will be compared between contact force-sensing guided or blinded strategy.

During 1-year follow up, patients who recurred AF or AT will be undergo second ablation procedure. In these patients, PV reconnection rate will be evaluated by a duodecapolar lasso circular mapping catheter. We would like to know whether PVs which have ablated with contact force-sensing information at index procedure have less reconnection than those which was ablated without contact force-sensing information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic paroxysmal atrial fibrillation (AF) who had failed with anti-arrhythmic agents.

Exclusion Criteria:

* Patients who had previous ablation for AF
* Patients with symptomatic persistent AF

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10-23 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Proportion of immediate PV isolation ratio after final ablation according to contact force-guided ablation, change of impedance, total ablation time, and procedure time according to contact force-guided strategy | Immediate after PV isolation (acute result)

SECONDARY OUTCOMES:
Proportion of PV reconnection according to contact force-guided ablation in patients with AF recurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Andrade JG, Monir G, Pollak SJ, Khairy P, Dubuc M, Roy D, Talajic M, Deyell M, Rivard L, Thibault B, Guerra PG, Nattel S, Macle L. Pulmonary vein isolation using "contact force" ablation: the effect on dormant conduction and long-term freedom from recurrent atrial fibrillation--a prospective study. Heart Rhythm. 2014 Nov;11(11):1919-24. doi: 10.1016/j.hrthm.2014.07.033. Epub 2014 Jul 25. PMID 25068575
- [Result] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Result] Marijon E, Fazaa S, Narayanan K, Guy-Moyat B, Bouzeman A, Providencia R, Treguer F, Combes N, Bortone A, Boveda S, Combes S, Albenque JP. Real-time contact force sensing for pulmonary vein isolation in the setting of paroxysmal atrial fibrillation: procedural and 1-year results. J Cardiovasc Electrophysiol. 2014 Feb;25(2):130-7. doi: 10.1111/jce.12303. Epub 2013 Nov 6. PMID 24433324
- [Result] Reichlin T, Knecht S, Lane C, Kuhne M, Nof E, Chopra N, Tadros TM, Reddy VY, Schaer B, John RM, Osswald S, Stevenson WG, Sticherling C, Michaud GF. Initial impedance decrease as an indicator of good catheter contact: insights from radiofrequency ablation with force sensing catheters. Heart Rhythm. 2014 Feb;11(2):194-201. doi: 10.1016/j.hrthm.2013.10.048. Epub 2013 Oct 28. PMID 24177370